CLINICAL TRIAL: NCT03009006
Title: Effect Of Combination of Calcium Hydroxide And Chlorhexidine Gel 2% as Intracanal Medication in Comparison to Calcium Hydroxide Paste as Intracanal Medication on Postoperative Pain And Bacterial Endotoxins in Necrotic Teeth:
Brief Title: Post Operative Pain and Level of Endotoxins With Calcium Hydroxide and Calcium Hydroxide Mixed With Chlorhexidine in Treating Necrotic Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Saadi Alarbeed, master candidate at endodontic department faculty of oral and dental medicine CU, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBC-CU-2016-10-147
Record Dates: First submitted 2016-12-30; First posted 2017-01-04 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Necrotic Pulp
Keywords: Calcium hydroxide intracanal medication; Ca(OH)2 intracanal medication; Chlorhexidene gel; CHX gel; Root canal treatment
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Calcium Hydroxide Mixed With Chlorhexidin (Experimental): efficacy of calcium hydroxide and 2 % chlorhexidine gel and combination of both on the anaerobic bacteria, It was clear from the study that calcium hydroxide had limited efficacy against facultative anaerobes, but effective against obligate anaerobes while chlorhexidine only and combination group were effective against all species of anaerobic bacteria.
  Interventions: Drug: Chlorhexidine 2% gel - Calcium Hydroxide Paste - Non-Setting
- Calcium Hydroxide (Experimental): The antimicrobial activity of calcium hydroxide Ca(OH)2 is related to the release of hydroxyl ions in an aqueous environment leading to damage in the bacterial cytoplasmic membrane, protein denaturation and DNA damage
  Interventions: Drug: Calcium Hydroxide Paste - Non-Setting
- Placebo (Placebo Comparator): Mechanical preparation without intracanal medications.
  Interventions: Drug: Chlorhexidine 2% gel - Calcium Hydroxide Paste - Non-Setting; Drug: Calcium Hydroxide Paste - Non-Setting

INTERVENTIONS:
Drug: Chlorhexidine 2% gel - Calcium Hydroxide Paste - Non-Setting — Calcium Hydroxide Mixed With Chlorhexidin efficacy of calcium hydroxide and 2 % chlorhexidine gel and combination of both on the anaerobic bacteria, It was clear from the study that calcium hydroxide had limited efficacy against facultative anaerobes, but effective against obligate anaerobes while chlorhexidine only and combination group were effective against all species of anaerobic bacteria
  Other Names: CHX gel; Ca(OH)2 paste
  Arms: Calcium Hydroxide Mixed With Chlorhexidin; Placebo
Drug: Calcium Hydroxide Paste - Non-Setting — Calcium Hydroxide The antimicrobial activity of calcium hydroxide Ca(OH)2 is related to the release of hydroxyl ions in an aqueous environment leading to damage in the bacterial cytoplasmic membrane, protein denaturation and DNA damage
  Other Names: Ca(OH)2 intracanal medication
  Arms: Calcium Hydroxide; Placebo

SUMMARY:
The aim of this prospective in vivo randomized clinical trial to evaluate influence of combination of calcium Hydroxide (CALCIPAST Paste, Poland) and chlorhexidine Gel 2% (Gluco-Chex 2%, Cerkamed, Poland) in comparison to calcium hydroxide paste (CALCIPAST Paste, Poland) as Intracanal Medication on post operative pain (incidence, degree, duration) and reduction of bacterial endotoxins (quantitative) after endodontic treatment in single rooted necrotic teeth.

According to the inclusion criteria the patients enrolled in the study and allocated randomly into three groups either combination of calcium hydroxide paste intracanal medication with 2% chlorhexidine gel. (group A) or calcium hydroxide paste intracanal medication only (group B) or mechanical preparation without intracanal medications (group C) the endodontic treatment is done at two visits.

The samples of endotoxin divided into three groups: after access (S1), after mechanical instrumentations (S2), after removal intracanal medication (S3), all samples taken by a sterile paper points introduced in the root canal for the working length for 60 seconds.

firstly the patient's medical and dental history is taken. the patients assign on informed consent. and then anaesthetized and access cavity performed and root canal preparation is done by Revo-s system then irrigation and intracanal medication placement inside to canal. the patient's record the post operative pain in sheet with NRS after 4, 24, 48 hours and 2 weeks after first visit. the operator will recall the patient to check the records

second visit After 2 weeks from application of ICM, rubber dam will be applied then removal of the temporary dressing, then a sterile paper point (S3) will be introduced into the canals after irrigation and removal of the remnants of the intracanal medicament with the saline solution.

* Removal of the paper sample to determine the endotoxin concentration.
* The canals will be obturated by single cone technique using gutta percha point tapered 0.4% (Gutta percha point, Revo-S MicroMega CO., LTD, France) corresponding to the final apical size of the file and the root canal sealer will be resin sealer (Adseal, META BIOMED CO., LTD, Korea).
* Pain will be assessed by numerical pain rating scale (NRS) after 14 days from the first visit (at the day of the Obturation) before the beginning of Obturation.

DETAILED DESCRIPTION:
Medical and dental history: diagnostic charts will be collected in a case report from by the investigators and confirmed for eligibility with the assistant supervisor.

Radiographic examination: preoperative radiographs will be taken to examine the tooth structure, caries detection, periapical status.

Clinical examination: intraoral examination include visual examination for caries, restorations, swelling, fistula, mobility, percussion were done.

Diagnostic criteria for necrotic tooth:

1. The patient marks moderate to severe pain on the numerical rating scale (NRS)a horizontal line of 11 marks and 10 intervals each takes number form 0 - 10 0 reading represents "no pain", 1- 3 readings represent "mild pain", 4- 6 readings represent "moderate pain", 7- 10 readings represent "severe pain".

   (recording baseline degree of pain preoperatively before initiating the endodontic treatment ) All step will done by operator.

   The measurement time will be at 4 hours, 24 hours, and 48 hours and after 14 days. (Day of Obturation)
2. The patient not responding to electric pulp tester at higher level than the contralateral tooth or the adjacent tooth if the contralateral one is missing.
3. Preoperative periapical x- ray film is done to detect any periapical changes.

Intervention:

Forty five patients will include were allocated by random or by chance to receive several clinical interventions and one of these interventions was control (Group A) where the patients did not receive any intracanal medication, (Group B) where the patients receive intracanal medication calcium hydroxide (CALCIPAST Paste, (Poland) and chlorhexidine 2 % gel. (Gluco-Chex 2%, Cerkamed, Poland), (Group C) calcium hydroxide paste only CALCIPAST Paste (Poland).

Procedure steps:

At the 1st appointment.

* Each patient will be given a numerical pain rating scale chart in order to rate his /her presenting pain as preoperative pain
* Anesthesia will be done with Carpule 3M™ ESPE™ Ubistesin™ Articaine HCI 4% & Adrenaline 1:100,000 3M Australia the tooth with decayed using a standard dental aspirating syringe.
* After diagnosis disinfecting the tooth surface by 30% H2O2 (Perfect Medical, Egypt) followed by 2.5% NaOCl inactivated with sodium thiosulfate (El Nasr CO. for pharmaceuticals and chemicals).
* Access cavity will do under rubber dam isolation and with Sterile burs for access cavity preparation with distilled water as a coolant and flaring will done by endo-z bur.
* If successful anesthesia occurs, working length will be determined with an apex locator (Root ZX, J.Morita, Irvine, California, USA.) then confirmed with intraoral periapical radiograph (Kodac Dental film, speed D, size 2, Carestream Health, Rochester, NY, USA) to confirm the length to be 0.5-1 mm shorter than radiographic apex.
* The first sample of endotoxin (S1) is taken by a sterile paper points after access cavity preparation and introduced in the root canal for the working length for 60 seconds.
* The sample is then placed in a pyrogenic free plastic tube and frozen to negative 200c for endotoxin determination by LAL test.
* Canal instrumentation will be done using NiTi rotary files system (Revo-S MicroMega, France) in an endodontic motor (X-Smart, Dentsply Maillefer, USA.) according to the manufacturer instructions to ensure adequate space for placement of the intracanal medicaments and proper removal of bacteria and debris, till size AS 35 file. The rotary files will be introduced inside the canal with EDTA gel (MD-Chelcream, META BIOMED CO., LTD, Korea) as lubricant.
* The irrigant solution will be NaOCl with concentration 2.5% for its tissue dissolving properties between each file and will be delivered by disposable plastic syringe.
* Another sample (S2) will be taken after the cleaning and shaping and before placing the intracanal medications by sterile paper point for endotoxin determination.
* The first group will be subjected to combined therapy of both calcium hydroxide intracanal medication CALCIPAST Paste (Poland), with 2% chlorhexidine gel intracanal medication (Gluco-Chex 2%, Cerkamed, Poland) after the cleaning and shaping for 2 weeks period.
* The second group will be subjected to calcium hydroxide intracanal medication alone for 2 weeks period after the cleaning and shaping. Calcium hydroxide will be in form of ready-made paste in a measured special syringe CALCIPAST (Poland).
* The third group will receive plain cotton with temporary filling without any intracanal medication.
* Placement of the intracanal medications by lentuolo spiral by low speed hand piece and condensed with paper points.
* Temporary filling is done by glass ionmer filling to ensure proper sealing with no leakage of any oral fluids inside the root canal, which may disturb the action of the intracanal medication.
* Pain will be assessed by numerical pain rating scale (NRS) will be given to each patient to complete a t home at the specified times at 4, 24, 48 hours after the first visit.

At the 2nd appointment:

* After 2 weeks from application of ICM, rubber dam will be applied then removal of the temporary dressing by following the previous infection control protocol, then a sterile paper point (S3) will be introduced into the canals after irrigation and removal of the remnants of the intracanal medicament with the saline solution.
* Removal of the paper sample to determine the endotoxin concentration.
* The canals will be obturated by single cone technique using gutta percha point tapered 0.4% (Gutta percha point, Revo-S MicroMega CO., LTD, France) corresponding to the final apical size of the file and the root canal sealer will be resin sealer (Adseal, META BIOMED CO., LTD, Korea).
* Pain will be assessed by numerical pain rating scale (NRS) after 14 days from the first visit (at the day of the Obturation) before the beginning of Obturation.

ELIGIBILITY:
Inclusion Criteria:

* Patients in Good Health(American Society Of Anaesthesiology Class II or higher).
* Adult patients from both genders older than 18-50 years old suffering from chronic periapical periodontitis with necrotic pulp.
* single rooted teeth (maxillary and mandibular).
* Patients who can understand numerical rating scale (NRS)
* Patients able to sign informed consent

Exclusion Criteria:

* Patients with Vital tooth.
* Patients having active pain in more than one tooth.
* Patients who had taken analgesics in 12 hours preceding the preparation.
* Any type of teeth with multi roots.
* Pulp hyperemia or any other conditions other than pulp necrosis like pulpitis or previously accessed teeth with temporary fillings and patients suffering from chronic disease (systemic diseases).
* Pregnant or mentally retarded patients.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2017-01-03; Primary Completion 2017-10 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | 4, 24, 48 hrs and 2 weeks after completion of treatment
  intensity of postoperative pain between visits by numerical Rating Scale (0- 10)

SECONDARY OUTCOMES:
bacterial endotoxins reductions | After access cavity, after mechanical preparation and after removal of intracanal medication (2 weeks after the first visit)
  bacterial endotoxins reduction will be assessed by ELISA technique.

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Elkhodary, Lecturer of Endodontics, Study Chair — Faculty of Oral and dental Medicine - Cairo University; Olfat Shaker, Professor, Principal Investigator — Faculty of Pharmacy - Cairo University.; Geraldine M. Ahmed, ass. professor, Study Director — Faculty of Oral and dental Medicine - Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh, Ripu Daman, et al.
- [Background] Walton RE, Holton IF Jr, Michelich R. Calcium hydroxide as an intracanal medication: effect on posttreatment pain. J Endod. 2003 Oct;29(10):627-9. doi: 10.1097/00004770-200310000-00003. PMID 14606782
- [Background] Siqueira JF Jr, Rocas IN. Clinical implications and microbiology of bacterial persistence after treatment procedures. J Endod. 2008 Nov;34(11):1291-1301.e3. doi: 10.1016/j.joen.2008.07.028. Epub 2008 Sep 17. PMID 18928835
- [Background] KAKEHASHI S, STANLEY HR, FITZGERALD RJ. THE EFFECTS OF SURGICAL EXPOSURES OF DENTAL PULPS IN GERM-FREE AND CONVENTIONAL LABORATORY RATS. Oral Surg Oral Med Oral Pathol. 1965 Sep;20:340-9. doi: 10.1016/0030-4220(65)90166-0. No abstract available. PMID 14342926
- [Background] Zehnder M. Root canal irrigants. J Endod. 2006 May;32(5):389-98. doi: 10.1016/j.joen.2005.09.014. PMID 16631834
- [Background] Gu LS, Kim JR, Ling J, Choi KK, Pashley DH, Tay FR. Review of contemporary irrigant agitation techniques and devices. J Endod. 2009 Jun;35(6):791-804. doi: 10.1016/j.joen.2009.03.010. PMID 19482174
- [Background] Cardoso MG, de Oliveira LD, Koga-Ito CY, Jorge AO. Effectiveness of ozonated water on Candida albicans, Enterococcus faecalis, and endotoxins in root canals. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2008 Mar;105(3):e85-91. doi: 10.1016/j.tripleo.2007.10.006. PMID 18280954
- [Background] Vianna ME, Horz HP, Conrads G, Zaia AA, Souza-Filho FJ, Gomes BP. Effect of root canal procedures on endotoxins and endodontic pathogens. Oral Microbiol Immunol. 2007 Dec;22(6):411-8. doi: 10.1111/j.1399-302X.2007.00379.x. PMID 17949345
- [Background] Nair PN, Sjogren U, Krey G, Kahnberg KE, Sundqvist G. Intraradicular bacteria and fungi in root-filled, asymptomatic human teeth with therapy-resistant periapical lesions: a long-term light and electron microscopic follow-up study. J Endod. 1990 Dec;16(12):580-8. doi: 10.1016/S0099-2399(07)80201-9. PMID 2094761
- [Background] Oliveira LD, Carvalho CA, Carvalho AS, Alves Jde S, Valera MC, Jorge AO. Efficacy of endodontic treatment for endotoxin reduction in primarily infected root canals and evaluation of cytotoxic effects. J Endod. 2012 Aug;38(8):1053-7. doi: 10.1016/j.joen.2012.04.015. Epub 2012 Jun 8. PMID 22794204
- [Background] Valera MC, da Rosa JA, Maekawa LE, de Oliveira LD, Carvalho CA, Koga-Ito CY, Jorge AO. Action of propolis and medications against Escherichia coli and endotoxin in root canals. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2010 Oct;110(4):e70-4. doi: 10.1016/j.tripleo.2010.01.029. PMID 20868987
- [Background] Bystrom A, Sundqvist G. The antibacterial action of sodium hypochlorite and EDTA in 60 cases of endodontic therapy. Int Endod J. 1985 Jan;18(1):35-40. doi: 10.1111/j.1365-2591.1985.tb00416.x. No abstract available. PMID 3922900
- [Background] Dametto FR, Ferraz CC, Gomes BP, Zaia AA, Teixeira FB, de Souza-Filho FJ. In vitro assessment of the immediate and prolonged antimicrobial action of chlorhexidine gel as an endodontic irrigant against Enterococcus faecalis. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2005 Jun;99(6):768-72. doi: 10.1016/j.tripleo.2004.08.026. PMID 15897866
- [Background] Estrela C, Sydney GB, Pesce HF, Felippe Junior O. Dentinal diffusion of hydroxyl ions of various calcium hydroxide pastes. Braz Dent J. 1995;6(1):5-9. PMID 8688650
- [Background] Gomes BP, Ferraz CC, Garrido FD, Rosalen PL, Zaia AA, Teixeira FB, de Souza-Filho FJ. Microbial susceptibility to calcium hydroxide pastes and their vehicles. J Endod. 2002 Nov;28(11):758-61. doi: 10.1097/00004770-200211000-00003. PMID 12470019
- [Background] Molander A, Reit C, Dahlen G, Kvist T. Microbiological status of root-filled teeth with apical periodontitis. Int Endod J. 1998 Jan;31(1):1-7. PMID 9823122
- [Background] Pinheiro ET, Gomes BP, Ferraz CC, Sousa EL, Teixeira FB, Souza-Filho FJ. Microorganisms from canals of root-filled teeth with periapical lesions. Int Endod J. 2003 Jan;36(1):1-11. doi: 10.1046/j.1365-2591.2003.00603.x. PMID 12656508
- [Background] Greenstein G, Berman C, Jaffin R. Chlorhexidine. An adjunct to periodontal therapy. J Periodontol. 1986 Jun;57(6):370-7. doi: 10.1902/jop.1986.57.6.370. PMID 3522851
- [Background] Ferraz CC, Gomes BP, Zaia AA, Teixeira FB, Souza-Filho FJ. In vitro assessment of the antimicrobial action and the mechanical ability of chlorhexidine gel as an endodontic irrigant. J Endod. 2001 Jul;27(7):452-5. doi: 10.1097/00004770-200107000-00004. PMID 11503994
- [Background] Siqueira JF Jr, de Uzeda M. Intracanal medicaments: evaluation of the antibacterial effects of chlorhexidine, metronidazole, and calcium hydroxide associated with three vehicles. J Endod. 1997 Mar;23(3):167-9. doi: 10.1016/S0099-2399(97)80268-3. PMID 9594757
- [Background] Sukawat C, Srisuwan T. A comparison of the antimicrobial efficacy of three calcium hydroxide formulations on human dentin infected with Enterococcus faecalis. J Endod. 2002 Feb;28(2):102-4. doi: 10.1097/00004770-200202000-00013. PMID 11833679
- [Background] Gomes BP, Souza SF, Ferraz CC, Teixeira FB, Zaia AA, Valdrighi L, Souza-Filho FJ. Effectiveness of 2% chlorhexidine gel and calcium hydroxide against Enterococcus faecalis in bovine root dentine in vitro. Int Endod J. 2003 Apr;36(4):267-75. doi: 10.1046/j.1365-2591.2003.00634.x. PMID 12702121
- [Background] Ohara P, Torabinejad M, Kettering JD. Antibacterial effects of various endodontic irrigants on selected anaerobic bacteria. Endod Dent Traumatol. 1993 Jun;9(3):95-100. doi: 10.1111/j.1600-9657.1993.tb00258.x. PMID 8243347
- [Background] Heling I, Steinberg D, Kenig S, Gavrilovich I, Sela MN, Friedman M. Efficacy of a sustained-release device containing chlorhexidine and Ca(OH)2 in preventing secondary infection of dentinal tubules. Int Endod J. 1992 Jan;25(1):20-4. doi: 10.1111/j.1365-2591.1992.tb00944.x. PMID 1399050
- [Background] Salzgeber RM, Brilliant JD. An in vivo evaluation of the penetration of an irrigating solution in root canals. J Endod. 1977 Oct;3(10):394-8. doi: 10.1016/S0099-2399(77)80172-6. No abstract available. PMID 270543
- [Background] Basrani B, Tjaderhane L, Santos JM, Pascon E, Grad H, Lawrence HP, Friedman S. Efficacy of chlorhexidine- and calcium hydroxide-containing medicaments against Enterococcus faecalis in vitro. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2003 Nov;96(5):618-24. doi: 10.1016/s1079-2104(03)00166-5. PMID 14600699
- [Background] Evans MD, Baumgartner JC, Khemaleelakul SU, Xia T. Efficacy of calcium hydroxide: chlorhexidine paste as an intracanal medication in bovine dentin. J Endod. 2003 May;29(5):338-9. doi: 10.1097/00004770-200305000-00005. PMID 12775006
- [Background] Estrela C, Holland R, Bernabe PF, de Souza V, Estrela CR. Antimicrobial potential of medicaments used in healing process in dogs' teeth with apical periodontitis. Braz Dent J. 2004;15(3):181-5. doi: 10.1590/s0103-64402004000300003. Epub 2005 Mar 18. PMID 15798819
- [Background] Schafer E, Bossmann K. Antimicrobial efficacy of chlorhexidine and two calcium hydroxide formulations against Enterococcus faecalis. J Endod. 2005 Jan;31(1):53-6. doi: 10.1097/01.don.0000134209.28874.1c. PMID 15614008
- [Background] Haenni S, Schmidlin PR, Mueller B, Sener B, Zehnder M. Chemical and antimicrobial properties of calcium hydroxide mixed with irrigating solutions. Int Endod J. 2003 Feb;36(2):100-5. doi: 10.1046/j.1365-2591.2003.00629.x. PMID 12657153
- [Background] Gomes BP, Vianna ME, Zaia AA, Almeida JF, Souza-Filho FJ, Ferraz CC. Chlorhexidine in endodontics. Braz Dent J. 2013;24(2):89-102. doi: 10.1590/0103-6440201302188. PMID 23780357
- [Background] Sinha N, Patil S, Dodwad PK, Patil AC, Singh B. Evaluation of antimicrobial efficacy of calcium hydroxide paste, chlorhexidine gel, and a combination of both as intracanal medicament: An in vivo comparative study. J Conserv Dent. 2013 Jan;16(1):65-70. doi: 10.4103/0972-0707.105302. PMID 23349580
- [Background] Sousa EL, Martinho FC, Nascimento GG, Leite FR, Gomes BP. Quantification of endotoxins in infected root canals and acute apical abscess exudates: monitoring the effectiveness of root canal procedures in the reduction of endotoxins. J Endod. 2014 Feb;40(2):177-81. doi: 10.1016/j.joen.2013.10.008. Epub 2013 Dec 10. PMID 24461400
- [Background] Adl A, Motamedifar M, Shams MS, Mirzaie A. Clinical investigation of the effect of calcium hydroxide intracanal dressing on bacterial lipopolysaccharide reduction from infected root canals. Aust Endod J. 2015 Apr;41(1):12-6. doi: 10.1111/aej.12054. Epub 2013 Dec 13. PMID 24330326
- [Background] Singh RD, Khatter R, Bal RK, Bal CS. Intracanal medications versus placebo in reducing postoperative endodontic pain--a double-blind randomized clinical trial. Braz Dent J. 2013;24(1):25-9. doi: 10.1590/0103-6440201302039. PMID 23657409
- [Background] Khattak, Yasir Khan, Shafqat Ali Shah, and Fayaz Alam.
- [Background] Asgary S, Eghbal MJ. Treatment outcomes of pulpotomy in permanent molars with irreversible pulpitis using biomaterials: a multi-center randomized controlled trial. Acta Odontol Scand. 2013 Jan;71(1):130-6. doi: 10.3109/00016357.2011.654251. Epub 2012 Feb 20. PMID 22339289